CLINICAL TRIAL: NCT05570864
Title: Artificial Intelligence Based Predictive Scoring System to Identify the Risk of Developing Cardiogenic Shock (CS) in Patients Suffering From Acute Coronary Syndrome (ACS)
Brief Title: Score TO Predict SHOCK - STOP SHOCK
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Premedix Academy (Other)
Responsible Party: Sponsor
Other Study IDs: 0012022
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Cardiogenic Shock; Acute Coronary Syndrome; Acute Myocardial Infarction
Keywords: cardiogenic shock; acute coronary syndrome; artificial intelligence; scoring system; machine learning; acute myocardial infarction
MeSH Terms: conditions — Shock, Cardiogenic; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group (with CS): A population of patients acquired from multiple national registries aged > 18 years, admitted for ACS without CS and proceeding to coronary angiography who developed cardiogenic shock (CS).
- Control group (without CS): A population of patients acquired from multiple national registries aged > 18 years, admitted for ACS without CS and proceeding to coronary angiography who did not develop cardiogenic shock (CS).

SUMMARY:
The goal of this international multicenter study is to develop a scoring system to identify the risk of developing cardiogenic shock (CS) in patients suffering from acute coronary syndrome (ACS) utilising artificial intelligence.

Study hypothesis:

A complex machine learning (ML) model utilising standard patient's admission data predicts the development of cardiogenic shock in patients suffering from acute myocardial infarction better than standard prediction models.

Study objectives:

The primary objective of this study is to further improve predictive parameters of #STOPSHOCK model for prediction of development of cardiogenic shock in patients suffering from acute myocardial infarction.

The secondary objective of this study is to develop a new predictive model for the development of cardiogenic shock in patients suffering from acute myocardial infarction based on larger combined cohort of patients utilising advanced ML algorithms, continuous model performance monitoring and continual learning.

DETAILED DESCRIPTION:
Background:

Cardiogenic shock is a serious life-threatening condition affecting almost 10% of patients suffering from acute coronary syndrome (ACS). When untreated, it can rapidly progress to collapse of circulation and sudden death. Despite recent improvements in diagnostic and treatment options, mortality remains incredibly high, reaching nearly 50%.

Currently available mechanical circulatory support devices can replace the function of the heart and/or lungs, thereby essentially eliminating the primary cause. However, cardiogenic shock is not only an isolated decrease in cardiac function but a rapidly progressing multiorgan dysfunction accompanied by severe cellular and metabolic abnormalities. The window for successful treatment is relatively narrow, and when missed, even the elimination of the underlying primary cause is not enough to reverse this vicious circle.

The ability to identify high-risk patients prior to the development of shock would allow to take pre-emptive measures, such as the implantation of mechanical circulatory support, and thus prevent the development of shock leading to improved survival.

Rationale:

The AI-based scoring system could aid in identifying high-risk patients prior to the development of cardiogenic shock. This would allow taking pre-emptive measures, implanting mechanical circulatory support, and thus prevent the development of shock, leading to improved survival.

For this purpose, a predictive scoring system STOP SHOCK (Score TO Predict SHOCK) was developed. This scoring system showed better prediction compared to standard models. STOP SHOCK was validated on an external cohort of patients with area under the curve (AUC) of 0.844 surpassing other externally validated cardiogenic shock (CS) models (e.g. ORBI score). Furthermore, this model is based on variables that are readily available at the first contact with patients and thus STOPSHOCK can be utilized in emergency room (ER) or ambulance even before catheterization.

ELIGIBILITY:
Inclusion criteria for study population:

1. Patients with at least one ICD9 diagnosis code:

   * 41000 - 41092: various versions of Acute myocardial infarction
   * 41189: Other acute and subacute forms of ischemic heart disease, other
   * 4139: Other and unspecified angina pectoris
2. Patients with at least one ICD9 diagnosis code:

   * 78551: Cardiogenic shock
   * 78550: Shock, unspecified
3. Patients with at least one ICD9 procedures codes:

   * 0066: Percutaneous transluminal coronary angioplasty [PTCA]
   * 3604: Intracoronary artery thrombolytic infusion
   * 3606: Insertion of non-drug-eluting coronary artery stent(s)
   * 3607: Insertion of drug-eluting coronary artery stent(s)
   * 3609: Other removal of coronary artery obstruction
   * 8855: Coronary arteriography using a single catheter
   * 8856: Coronary arteriography using two catheters
   * 8857: Other and unspecified coronary arteriography
   * 3722: Left heart cardiac catheterization
   * 3723: Combined right and left heart cardiac catheterization

Inclusion criteria for control group:

1. Patients with at least one ICD9 diagnosis code:

   * 41000 - 41092: various versions of Acute myocardial infarction
   * 41189: Other acute and subacute forms of ischemic heart disease, other
   * 4139: Other and unspecified angina pectoris
2. Patients with at least one of the ICD9 procedures codes:

   * 0066: Percutaneous transluminal coronary angioplasty [PTCA]
   * 3604: Intracoronary artery thrombolytic infusion
   * 3606: Insertion of non-drug-eluting coronary artery stent(s)
   * 3607: Insertion of drug-eluting coronary artery stent(s)
   * 3609: Other removal of coronary artery obstruction
   * 8855: Coronary arteriography using a single catheter
   * 8856: Coronary arteriography using two catheters
   * 8857: Other and unspecified coronary arteriography
   * 3722: Left heart cardiac catheterization
   * 3723: Combined right and left heart cardiac catheterization

Exclusion criteria for control group:

1. Patients without ICD9 diagnosis codes:

* 78551: Cardiogenic shock
* 78550: Shock, unspecified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a combined population of patients who suffered acute myocardial infarction recorded in national registries from several countries. An estimated 30 to 50000 new patients will be added from multiple registries to to improve the existing primary STOP SHOCK model. The incidence of cardiogenic shock in this group of patients is estimated to be 10% which would constitute the shock patient group, the rest of the patients will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Development of cardiogenic shock | Up to 72 hours
  Development of cardiogenic shock (CS) in patients suffering from acute coronary syndrome (ACS)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Böhm, MD, PhD, MBA, FESC, FJCS, Principal Investigator — Premedix Academy, Medena 18, 81102 Bratislava, Slovakia
Locations (1):
- Premedix Academy, Bratislava, Slovakia

REFERENCES:
- See also: STOP SHOCK website — https://stopshock.org/